CLINICAL TRIAL: NCT02086669
Title: Randomized Study to Compare Pneumatic Dilatation With Surgical Myotomy for Treatment of Achalasia - Long Term Follow up
Brief Title: Pneumatic Dilatation or Surgical Myotomy for Achalasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Lars Lundell, Professor, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S500-00
Record Dates: First submitted 2014-03-03; First posted 2014-03-13 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Achalasia
MeSH Terms: conditions — Esophageal Achalasia | interventions — Heller Myotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pneumatic dilatation (Experimental): Repetitive pneumatic dilatation as the initial treatment followed by repetitive dilatation in case of dysphagia recurrence.
  Interventions: Procedure: Pneumatic dilatation
- Surgical myotomy (Active Comparator): Laparoscopic myotomy and subsequent follow up.
  Interventions: Procedure: Laparoscopic myotomy

INTERVENTIONS:
Procedure: Pneumatic dilatation
  Arms: Pneumatic dilatation
Procedure: Laparoscopic myotomy
  Arms: Surgical myotomy

SUMMARY:
Patients with newly diagnosed achalasia have been submitted to either treatment with pneumatic dilatation or surgical myotomy. Minimal follow up five years.

DETAILED DESCRIPTION:
Patients with newly diagnosed achalasia have been submitted to either treatment with pneumatic dilatation or surgical myotomy. Minimal follow up five years.

During follow up patients have been interviewed with regular intervals, by use validated questionnaires. The level of symptom control has been assessed as well as the scoring cumulative incidence of treatment failures.

Health Related Quality of Life (HRQL) has been regularly checked.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed achalasia
* Age 18-80 years
* Informed consent

Exclusion Criteria:

* Previous treatment for achalasia.
* Stage IV achalasia.
* Unwillingness to participate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2000-01; Primary Completion 2009-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Treatment failures | At least five years after intervention
  Treatment failure is defined as a Composite variabel containing a number of different Clinically relevant outcomes.

SECONDARY OUTCOMES:
Dysphagia scoring | At least five years after intervention
  Dysphagia score according to standardized, validated scoring system.
Health Related Quality of Life | At least five years after intervention.
  Universally adopted and validated instruments are used.
Direct medical costs. | At least five years after intervention.
  Charges for the average hospital in respective countries.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Lundell, Professor, Study Chair — Karolinska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Derived] Persson J, Johnsson E, Kostic S, Lundell L, Smedh U. Treatment of achalasia with laparoscopic myotomy or pneumatic dilatation: long-term results of a prospective, randomized study. World J Surg. 2015 Mar;39(3):713-20. doi: 10.1007/s00268-014-2869-4. PMID 25409838